CLINICAL TRIAL: NCT04613609
Title: Vaporized Nicotine and Autonomic Control
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michigan Technological University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: M1747
Record Dates: First submitted 2020-10-15; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Electronic Cigarette Use
Keywords: E-cigarette; Autonomic Control; Muscle Sympathetic Nerve Activity
MeSH Terms: conditions — Vaping | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Repeated Measures
Who Masked: Participant
Masking Description: Participants were not informed if they were to receive nicotine or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): E-cigarette containing no nicotine.
  Interventions: Device: Electronic Cigarette without nicotine
- Nicotine (Active Comparator): E-cigarette containing nicotine
  Interventions: Device: Electronic Cigarette containing nicotine

INTERVENTIONS:
Device: Electronic Cigarette containing nicotine — Non-smokers used an electronic cigarette containing nicotine
  Other Names: JUUL (brand name)
  Arms: Nicotine
Device: Electronic Cigarette without nicotine — Non-smokers used an electronic cigarette without nicotine
  Other Names: Smok (brand name)
  Arms: Placebo

SUMMARY:
E-cigarettes are marketed as an alternative to smoking for those who want to decrease the health risks of tobacco. Tobacco cigarettes increase heart rate (HR) and arterial pressure, while reducing muscle sympathetic nerve activity (MSNA) through sympathetic baroreflex inhibition. The acute effects of e-cigarettes on arterial pressure and MSNA have not been reported: our purpose was to clarify this issue. Using a randomized crossover design, participants inhaled on a JUUL containing nicotine (59 mg/ml) and a similar placebo e-cigarette (0 mg/ml).

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Individuals with a history of hyperthyroidism
* Women currently taking oral contraceptives, are pregnant or breast-feeding, or trying to become pregnant
* Individuals currently taking prescription drugs.
* Individuals with respiratory illnesses (e.g., asthma, chronic obstructive pulmonary disease, reactive airway disease, etc.)
* Individuals with hypertension (systolic >130 and/or diastolic > 80).
* Individuals with a history of tobacco or vaporized nicotine use.
* Individuals who have been diagnosed with diabetes
* Individuals who are under the age of 18 or over the age of 40

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure (measured from the finger) | Experiments were separated by one month. Beat-to-beat arterial pressure was recorded for ten minutes at rest, during ten minutes of e-cigarette use, and for ten minutes during recovery. The last 5 minutes of each section were averaged.
  Effects of electronic cigarettes on both systolic and diastolic arterial pressure.
Muscle sympathetic nerve activity (measured with the microneurography technique) | Experiments were separated by one month. MSNA was recorded for ten minutes at rest, during ten minutes of e-cigarette use, and for ten minutes during recovery. The last 5 minutes of each section were averaged.
  Effects of electronic cigarettes on muscle sympathetic nerve activity (MSNA)

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Technological University, Houghton, Michigan, United States